CLINICAL TRIAL: NCT01159613
Title: Do Low HDL Levels Predict Treatment Outcome in Patients With Chronic Hepatitis C Viral Infection?
Brief Title: Do Low High Density Lipoprotein (HDL) Levels Predict Treatment Outcome in Patients With Chronic Hepatitis C Viral Infection?
Status: Completed | Type: Observational
Sponsor: Ziv Hospital (Other Government)
Collaborators: Hillel Yafe MC Hadera (Unknown)
Responsible Party: Liver Clinic, Ziv medical center
Other Study IDs: HDL + HCV
Record Dates: First submitted 2010-07-08; First posted 2010-07-09 (Estimated); Last update posted 2010-07-09 (Estimated); Status verified 2010-07

CONDITIONS: Chronic Hepatitis C Viral Infection
Keywords: SVR; Cholesterol level; fibrosis score; HDL

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Non Responders: Non Responders
  Interventions: Other: Non Responders
- RESPONDERS
  Interventions: Other: Responders

INTERVENTIONS:
Other: Responders — Responders
  Groups: RESPONDERS
Other: Non Responders — Non Responders
  Groups: Non Responders

SUMMARY:
The working hypothesis is that the low HDL serum level predict favorable response to anti viral treatment in chronic HCV (genotype 1) viral infection. This might be used to improve the rate of sustained virologic response.

DETAILED DESCRIPTION:
Lipoproteins are closely connected to the process of hepatitis C virus (HCV) infection. Metabolic syndrome predicts negative treatment outcome in HCV infection.

Aim: to assess the association between lipids components of the metabolic syndrome and sustained viral response (SVR).

ELIGIBILITY:
Inclusion Criteria:

* Chronic HCV genotype 1 naive patients

Exclusion Criteria:

* Co infection with HBV, HIV, HDV
* Decompensated liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: chronic HCV genotype 1 naïve patients
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2008-04; Primary Completion 2008-10 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
sustained viral response | 72 weeks
  achieving SVR

CONTACTS AND LOCATIONS:
Locations (1):
- Ziv medical center liver unit, Safed, Israel, Israel